CLINICAL TRIAL: NCT00000178
Title: Multicenter Trial of Prednisone in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0002; 3U01AG010483-08S2 (NIH)
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Prednisone; Anti-inflammatory agents
MeSH Terms: conditions — Alzheimer Disease | interventions — Prednisone

INTERVENTIONS:
Drug: Prednisone

SUMMARY:
This is a randomized placebo controlled, double blind study. Patients who meet eligibility criteria and decide to participate in the study will be randomly assigned to receive either drug treatment or a placebo. Neither the patients nor the participating investigators will know who is receiving the drugs and who is receiving the placebo. Participation involves 15 outpatient clinic visits over a 68 week period. Patients take study medication at varying doses (the maximum dose is 20 mg daily), along with calcium and vitamin supplements.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Alzheimer's disease who are in stable medical condition

Exclusion Criteria:

* Patients with diabetes or severe osteoporosis

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Leon Thal, MD., Principal Investigator — University of California, San Diego
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University Alzheimer's Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Burke Medical Research Institute, White Plains, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Dallas, Texas

REFERENCES:
- [Result] Aisen PS, Davis KL, Berg JD, Schafer K, Campbell K, Thomas RG, Weiner MF, Farlow MR, Sano M, Grundman M, Thal LJ. A randomized controlled trial of prednisone in Alzheimer's disease. Alzheimer's Disease Cooperative Study. Neurology. 2000 Feb 8;54(3):588-93. doi: 10.1212/wnl.54.3.588. PMID 10680787
- See also: The Alzheimer's Disease Education and Referral (ADEAR) Center is a service of the National Institute on Aging (NIA). — http://www.alzheimers.org